CLINICAL TRIAL: NCT01852227
Title: ADAPT A Direct Aspiration, First Pass Technique for the Endovascular Treatment of Stroke
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: State University of New York - Downstate Medical Center (Other); Stony Brook University (Other); Swedish Medical Center (Other); Vanderbilt University (Other); West Virginia University (Other)
Responsible Party: Sponsor
Other Study IDs: PRO23524
Record Dates: First submitted 2013-04-23; First posted 2013-05-13 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-08

CONDITIONS: Stroke Technique

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In collaboration with the Neurointerventional programs at state university of new york Buffalo, state university of new york Stonybrook, Swedish Medical Center, Erlanger Health System, Vanderbilt University, and West Virginia University School of Medicine, the investigators aim to prospectively collect experiences where direct aspiration as a first pass technique is used for thrombectomy procedures.

The investigators also want to compare specific characteristics from these cases to other stroke cases where traditional thrombectomy devices were used.

DETAILED DESCRIPTION:
Traditionally, at a physician's discretion, first pass attempts at thrombectomy procedures are performed with any number of FDA cleared catheters, guide wires, and devices designed for efficient removal of clot within an intracranial vessel. Among institutions involved in this case study, the latest devices are readily available and fully support standard treatment paradigms.

However, several cases, recently completed, using only large bore catheter and aspiration have anecdotally demonstrated a superior ability to remove clot from vessels, restoring blood flow to the affected vessel and brain tissue. In these limited number of cases, full restoration of blood flow has been achieved. While this combination of approved devices is minimalistic, the efficiency of the procedure, rapid technical success, and relative simplicity of the approach is unique and should be thoroughly reviewed and possibly prepared for publication.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were treated with direct aspiration as a first pass choice or treated with a stent retriever will be included.

Exclusion Criteria:

* Patients not treated with either direct aspiration as a first pass, or stent retriever will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a chart review of clinical data for patients who have been treated for stroke with either direct aspiration or stent retrievers. This review will be conducted at MUSC and SUNY Buffalo, SUNY Stonybrook, Swedish Medical Center, Vanderbilt University, Erlanger Health System, and West Virginia University School of Medicine. Each participating group will submit for approval at their individual institution.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Discharge national institutes of health stroke scale (NIHSS) | approximately 7 days after index stroke
  a national institutes of health stroke scale (NIHSS) will be obtained at the time of the each patient's discharge or approximately 7 days

SECONDARY OUTCOMES:
90 day modified Rankin Score (mRS) | 90 days after procedure
  90 days after procedure each patient's modified Rankin Score will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Aquilla Turk, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States